CLINICAL TRIAL: NCT03392909
Title: Restoration of Full-Length Type VII Collagen in RDEB Patients With Nonsense Mutations After Intravenous Gentamicin Treatment
Brief Title: Intravenous Gentamicin Therapy for Recessive Dystrophic Epidermolysis Bullosa (RDEB)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, David Woodley, Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-17-00995
Record Dates: First submitted 2018-01-02; First posted 2018-01-08 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Recessive Dystrophic Epidermolysis Bullosa
Keywords: Nonsense Mutations
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica | interventions — Gentamicins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intravenous Gentamicin (Experimental): Intravenous gentamicin (7.5 mgs/kg) daily for for either 14 days and then stopped or twice weekly for three months and then stopped.
  Interventions: Drug: Gentamicin

INTERVENTIONS:
Drug: Gentamicin — Short-term intravenous gentamicin therapy should have the advantage of treating all of the patient's multiple skin wounds simultaneously. Six patients (three adults and 3 children) will receive intravenous gentamicin (7.5 mgs/kg) daily for 14 days and then stopped. Three adult patients will receive intravenous gentamicin (7.5mg/kg) biweekly for three months and then stopped.
  Other Names: Gentamicin Sulfate

SUMMARY:
Recessive dystrophic epidermolysis bullosa (RDEB) is an incurable, devastating, inherited skin disease caused by mutations in the COL7A1 gene that encodes for type VII collagen (C7), the major component of anchoring fibrils (AFs), structures that mediate epidermal-dermal adherence. Thirty percent of RDEB patients have nonsense mutations. The investigators recently demonstrated in 5 such patients that intradermal and topical gentamicin induced "read-through" of their nonsense mutations and created robust and sustained new C7 and AFs at the dermal-epidermal junction (DEJ) of their skin and also stimulated wound closure and reduced new blister formation. No untoward side effects occurred. Herein, the investigators propose evaluating the safety and efficacy of intravenous gentamicin in these patients. In theory, this intravenous administration has the possibility of treating simultaneously all of the patients' skin wounds. The milestones will be increased C7 and AFs in the patients' DEJ, improved EB Disease Activity Scores, and absence of gentamicin side effects.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 7 and up can participate in the 14 day IV gentamicin trial. Male or female, aged 18 and up can participate in the 3 month IV gentamicin trial.
* Been diagnosed with recessive dystrophic epidermolysis bullosa (RDEB) and with a nonsense mutation in the COL7A1 gene.
* Immunofluorescence evaluation of skin biopsies reveals absence or decreased intensity of C7 expression at their DEJ (dermal epidermal junction) compared with normal human skin biopsies.
* Cultured fibroblasts from patient skin synthesize and secrete full-length, 290kDa C7 alpha chains in the presence of supplemented gentamicin (400 μg/ml in culture).
* Ability to sit or lie down for over 30 minutes for IV infusions. For those in the 3 month trial, to be willing to continue treatment at home under the supervision of licensed and trained infusion nurses.

Exclusion Criteria:

* Recent exposure to gentamicin within the past 6 weeks.
* Pre-existing known auditory impairment.
* Pre-existing known renal impairment.
* Pre-existing known allergies to aminoglycosides or sulfate compounds.
* Pregnancy or lactation
* Current use of medications with known ototoxicity or nephrotoxicity.
* Current enrollment in another experimental clinical trial involving systemic treatment with C7 or C7 producing products for the treatment of RDEB.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2018-07-05 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Full-length type VII collagen expression | 6 months
  Increased expression of full-length type VII collagen as assessed by immunofluorescence
Generation of anchoring fibrils | 6 months
  Generation of new anchoring fibrils as assessed by immuno-electron microscopy
Absence of gentamicin side effects | 6 months
  Absence of gentamicin side effects, especially the detection of any ototoxicity or nephrotoxicity

SECONDARY OUTCOMES:
Improved Disease Activity scores | 6 months
  Improved epidermolysis bullosa Disease Activity scores
Improved Quality of Life score | 6 months
  Improved Quality of Life score

CONTACTS AND LOCATIONS:
Overall Officials: David T. Woodley, MD, Principal Investigator — Professor, University of Southern California; Mei Chen, Ph.D, Principal Investigator — Professor, University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No